CLINICAL TRIAL: NCT04358367
Title: Intravenous Dexmedetomidine Reduces Hypotension and Epigastric Pain in Cesarean Section Under Spinal Anesthesia: A Randomized Clinical Study
Brief Title: Intravenous Dexmedetomidine in Cesarean Section Under Spinal Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 01041620
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-04

CONDITIONS: Cesarean Section Complications
Keywords: dexmedetomidine; spinal anesthesia; cesarean section; epigastric pain
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): spinal anesthesia and intravenous dexmedetomidine(1µg/kg)
  Interventions: Drug: Dexmedetomidine Injectable Product
- Saline (Placebo Comparator): spinal anesthesia and placebo (saline).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine Injectable Product — Spinal anesthesia and intravenous dexmedetomidine (1μg/kg). The administrated drugs were slowly injected intravenously over 10 minutes then intrathecal block was achieved using 2-2.2 ml of hyperbaric bupivacaine (10 -12.5 mg) introduced at L3/4 or L4/5 interspace.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Saline — Spinal anesthesia and intravenous saline. The administrated drugs were slowly injected intravenously over 10 minutes then intrathecal block was achieved using 2-2.2 ml of hyperbaric bupivacaine (10 -12.5 mg) introduced at L3/4 or L4/5 interspace.
  Other Names: saline solution
  Arms: Saline

SUMMARY:
The present study hypothesized that intravenous dexmedetomidine use during spinal anesthesia for cesarean section has a beneficial influence on hemodynamic stability and epigastric pain together with satisfactory analgesic effects and excellent safety profile for the mother and the newborn.

DETAILED DESCRIPTION:
Background and aim: Hypotension and epigastric pain are commonly encountered during spinal anesthesia for cesarean section. Dexmedetomidine (DEX) is a highly selective α 2-adrenergic agonist. Its effects entail sympatholytic, sedative, anesthetic, and analgesic actions. The present randomized study aimed to evaluate the effect of intravenous DEX administration on the hemodynamic parameters and epigastric pain in women subjected to cesarean section.

Patients and Methods: This study is a randomized double-blinded controlled trial. Seventy patients were randomly assigned to one of two interventional groups: one group received spinal anesthesia and intravenous DEX (1µg/kg) and the other group received spinal anesthesia and placebo (saline). The administrated drugs were slowly injected intravenously over 10 minutes then intrathecal block was achieved using 2-2.2 ml of hyperbaric bupivacaine (10 -12.5 mg) introduced at L3/4 or L4/5 interspace. Primary Outcome parameters included frequency of hypotension episodes, frequency of ephedrine doses needed, sedation score and epigastric pain episodes. Secondary outcomes included time to onset of sensory and motor blocks, duration of sensory and motor blocks, operative duration, time needed to request of rescue analgesia, level of intrathecal block, and neonatal Apgar score at 1 and 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Full-term pregnancy and American Society of Anesthesiologists (ASA) physical status I/II in women scheduled for elective cesarean section

Exclusion Criteria:

* Severe hepatic or renal disease
* Severe cardiopulmonary disease
* Thyroid disorders multiple allergies prematurity
* Known fatal abnormality
* Known chronic gastrointestinal problems with epigastric pain e.g. peptic ulcer and reflux esophagitis.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2019-05-19 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
hypotension | up to 48 hours postoperative
  systolic blood pressure < 90 mmHg
ephedrine use | up to 48 hours postoperative
  frequency of ephedrine doses needed
sedation | up to 48 hours postoperative
  sedation score
epigastric pain | up to 48 hours postoperative
  Pain in the epigastric region assessed by Visual Analog Scale

SECONDARY OUTCOMES:
sensory and motor blocks | Intraoperative
  time to onset of sensory and motor blocks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elsawy, MD, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Azhar University Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No